CLINICAL TRIAL: NCT03843021
Title: Understanding and Addressing Variation in Healthcare-Associated Infections After Durable Ventricular Assist Device Therapy: Organizational: Aim 1 Survey
Brief Title: Ventricular Assist Device (VAD) Infection Prevention Survey
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Donald Likosky, Principal Investigator, University of Michigan
Other Study IDs: HUM00157335
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure; Healthcare Associated Infection; Ventricular Assist Device
MeSH Terms: conditions — Heart Failure; Cross Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VAD Healthcare Providers: Adult healthcare providers of VAD therapy recipients.
  Interventions: Other: VAD Infection Prevention Survey

INTERVENTIONS:
Other: VAD Infection Prevention Survey — Healthcare providers caring for VAD Therapy recipients will answer questions regarding processes of care at their institutions.

SUMMARY:
Annually, more than 250,000 patients in the U.S. with end-stage heart failure stand to benefit from ventricular assist device (VAD) therapy. 60% of patients develop a healthcare-associated infection (HAI) within 90-days of implantation. The investigators long term goal is to develop and subsequently promote wide-scale adoption of evidence-based HAI prevention practices following durable VAD implantation.

This will be done by addressing the following aims:

Aim 1. Identify determinants of center-level variability in HAI rates. Aim 2. Develop a comprehensive understanding of barriers and facilitators for achieving low center HAI rates.

Aim 3. Develop, iteratively enhance, and disseminate a best practices toolkit for preventing HAIs that accommodates various center contexts.

The investigators will use a focused survey of U.S. VAD centers to identify determinants of center variation in 90-day HAI rates:

* Process Factors (e.g., intranasal mupirocin),
* Provider Factors (e.g., surgeon technique),
* Device Factors (e.g., centrifugal vs. axial),
* Center Factors (e.g., provider communication).

Understanding the barriers and facilitators within individual centers for maximizing adoption of prevention measures would serve as the foundation for targeted improvement strategies. Without this knowledge, evidence-based, action-oriented recommendations will have limited local adoption and ultimately effectiveness in preventing HAIs after VAD implantation.

DETAILED DESCRIPTION:
Annually, more than 250,000 patients in the U.S. with end-stage heart failure stand to benefit from ventricular assist device (VAD) therapy. Despite VADs providing long-term "durable" support, this therapy is associated with substantial risk (50% mortality at 4 years) and expense ($179,000 for inpatient services). Additionally, 60% of patients develop a healthcare-associated infection (HAI) within 90-days of implantation. Broad adoption of durable VAD therapy is hindered in part by HAIs, given associated sequelae (6-fold increased risk of 1-year mortality) and costs ($264,000 - $869,000 per patient). It is critical to determine how best to prevent HAIs in order to maximize the benefit of VAD therapy. While several studies have reported variation in HAI rates across centers after complex cardiac surgery, less is known in the setting of durable VADs. The average 90-day HAI rate after VAD implantation is as high as 19 events per 100 patient-months and varies (25th - 75th percentile, 9-23) across centers. While some argue that centers with lower HAI rates select healthier patients, others counter that improved practices (e.g., standardizing empirical and targeted antimicrobial therapy) or enhanced provider teamwork are more predictive of improved outcomes.

While evidence-based HAI prevention guidelines and implementation tools (e.g., checklists) exist, these approaches are not comprehensive (e.g., neglecting device-specific determinants) or customizable to local context, thus limiting usability, adoption, and likelihood of significant effectiveness for preventing HAIs. Understanding the barriers and facilitators within individual centers for maximizing adoption of prevention measures would serve as the foundation for targeted improvement strategies. Without this knowledge, evidence-based, action-oriented recommendations will have limited local adoption and ultimately effectiveness in preventing HAIs after VAD implantation.

The investigators long-term goal is to develop and subsequently promote wide-scale adoption of evidence-based HAI prevention practices following durable VAD implantation. The objective of this proposal is to identify prevention recommendations for the most significant HAIs after VAD implantation. To achieve this objective, the investigators will undertake a mixed methods study of adult patients receiving VADs in the U.S. from 2009 - 2017 and develop a modular toolkit of evidence-based recommendations. To determine best practices for preventing HAIs, the investigators will examine center-level differences in HAI rates to identify strategies used by centers with low rates, and potential barriers among centers with high rates.

ELIGIBILITY:
Inclusion Criteria:

Healthcare providers involved in the medical management of a Ventricular Assist Device (VAD) recipient during the peri-operative period, including those with the following roles: surgeons, cardiologists and VAD coordinators

Exclusion Criteria:

Healthcare providers not caring for VAD recipient patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare providers involved in the medical management of a Ventricular Assist Device (VAD) recipient during the peri-operative period, specifically surgeons, cardiologist, VAD coordinators.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
An organization's use of practices associated with center HAI rates. | March 2019 - March 2020
  We will use a survey to identify a center's use of practices that may explain their center's HAI rate

CONTACTS AND LOCATIONS:
Overall Officials: Donald S Likosky, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing individual participant data